CLINICAL TRIAL: NCT00757003
Title: A Clinical Study of the TAG Thoracic Endoprosthesis in the Treatment of Thoracic Aortic Diseases for Non-Surgical Candidates Under the Physician Sponsored IDE.
Brief Title: To Evaluate the Safety and Efficacy for GORE TAG Thoracic Endoprosthesis in the Treatment of Thoracic Aortic Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Daniel Yung-Ho Sze, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-09112008-1299; 13335 (SQL 73498) (Other: Stanford University)
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Aneurysm, Dissecting; Aortic Aneurysm, Thoracic
MeSH Terms: conditions — Aortic Dissection; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm - Placement of TAG device (Experimental): A TAG device will be used to repair the pathology in the thoracic aorta
  Interventions: Device: Endovascular Stent-graft repair of descending thoracic aorta

INTERVENTIONS:
Device: Endovascular Stent-graft repair of descending thoracic aorta — A TAG device will be used to repair the pathology in the thoracic aorta

SUMMARY:
PURPOSE OF RESEARCH:

Endovascular stent-graft repair of aortic pathologies is a minimally-invasive alternative to open surgery that may decrease morbidity and mortality, particularly in high risk patients. Optimal patient selection, based on pathology and anatomy, is being defined. Technically successful implantation requires adequate assessment of pathology and anatomy, and development and execution of novel and delicate procedures that resolve the pathology while minimizing morbidity and mortality.

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

There will be a maximum of 100 patients treated with the new device. You will be evaluated by your doctor to determine if you are able to participate in this research study. This evaluation will include reviewing your medical history, a physical examination, and special x-rays. These special x-rays are called CT scans and angiograms. Your doctor will explain what tests you will have done. A CT scan is a special x-ray that allows your doctor to see the size and shape of your aorta and your arteries. An angiogram uses a catheter (a hollow tube) that is placed into your arteries. Both tests use dye that can be seen on x-rays to see how the blood flows through your aorta and the surrounding arteries; for the CT scan it will be injected into a vein, and for the angiogram it is injected through the catheter into your arteries. These tests would be conducted whether or not you were participating in this research study. Your doctor will use this type of testing to determine if you are eligible to participate in this research study and as part of your follow-up care. Currently there are two aortic stent grafts manufactured by W.L. Gore & Associates that are approved by the FDA for experimental use. Your doctor will determine which device is more appropriate to treat your condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be poor or high risk open surgical candidates.
2. Thoracic aortic disease deemed to warrant exclusion in order to prevent rupture or extension including dissection and transection.
3. Anatomy meets TAG Endoprosthesis specification criteria.
4. Minimum 2 cm non-aneurysmal segment proximal and distal to the aneurysm

   * <60 angle in the aortic arch may require additional length of non-aneurysmal segment is the arch is included in the treatment segment.
5. Ability to comply with protocol requirements including follow-up.
6. Signed Informed Consent

Exclusion Criteria:

1. >4mm aortic taper and inability to use devices of different diameters, to compensate for the taper, in the treatment area of the aorta.
2. Significant thrombus at the proximal or distal implantation sites.
3. Planned occlusion of the left carotid or celiac arteries, unless supplemental conduit or alternate perfusion routes for end organ(s) provided.
4. Degenerative connective tissue disease, e.g. Marfan's or Ehler's Danlos Syndrome, unless the proximal and distal implantation sites of the TAG Endoprosthesis are located with in previous surgical grafts.

6. Female of child bearing age with positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2001-10; Primary Completion 2013-07 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Yung-Ho Sze, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data is made available upon request to colleagues conducting similar studies throughout the US.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment October 2000 - November 2007. Patients presenting or transferred to Stanford University Medical Center with thoracic aortic pathology deemed prohibitively high risk for open surgical repair.
Groups:
- Treatment Arm - Placement of TAG Device: Endovascular Stent-graft repair of descending thoracic aorta: A TAG device will be used to repair the pathology in the thoracic aorta. Pathology may include aneurysm, dissection, penetrating ulcer, pseudoaneurysm, false aneurysm, transection, mycotic aneurysm.
Period: Overall Study
Arm/Group | Treatment Arm - Placement of TAG Device
Started | 100
Completed | 51
Not Completed | 49
Not completed — Death | 33
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal by Subject | 4
Not completed — Surgically explanted | 2
Not completed — Not implanted | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm - Placement of TAG Device
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (17.4)
Gender [Count of Participants; unit: Participants]
  Female | 31
  Male | 69

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Technically Successful Implant
Description: The percentage of participants with technically successful implantation as assessed by the investigator is reported.
Time Frame: Day 0 to Day 30
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm - Placement of TAG Device
Number analyzed (Participants) | 100
percentage of participants | 99.0

2. Secondary Outcome: Count of Participants Experiencing at Least One Endoleak Following Procedure
Description: Endoleak is persistent blood flow in the aneurysm sac.
Time Frame: Up to 60 months following procedure
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm - Placement of TAG Device: A TAG device will be placed in the Aorta to treat the AAA. A TAG device will be used to repair the aneurysm in the thoracic aorta
  Endovascular Stent-graft repair of descending thoracic aorta: A TAG device will be used to repair the aneurysm in the thoracic aorta
Arm/Group | Treatment Arm - Placement of TAG Device
Number analyzed (Participants) | 100
Participants | 32

3. Secondary Outcome: Overall Survival
Description: Overall survival is reported as the count of participants alive 60 months following implant procedure.
Time Frame: 60 months
Population: 9 lost to followup, 4 withdrew, 2 explanted, 1 never implanted, all excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm - Placement of TAG Device
Number analyzed (Participants) | 84
Participants | 51

ADVERSE EVENTS:
Arm/Group | Treatment Arm - Placement of TAG Device
Serious Adverse Events (participants affected / at risk) | 43/100
Other Adverse Events (participants affected / at risk) | 16/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm - Placement of TAG Device (N=100)
Atelectasis/Pneumonia (Respiratory, thoracic and mediastinal disorders) | 28 (28)
cardiac arrhythmia (Cardiac disorders) | 21 (21)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 (13)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 (12)
change in mental status (Nervous system disorders) | 11 (11)
cerebrovascular accident (Nervous system disorders) | 8 (8)
renal failure (Renal and urinary disorders) | 9 (9)
renal insufficiency (Renal and urinary disorders) | 7 (7)
procedural hemorrhage (Surgical and medical procedures) | 12 (12)
paraplegia/paraparesis (Nervous system disorders) | 1 (1)
type I endoleak (Surgical and medical procedures) | 13 (13)
type II endoleak (Surgical and medical procedures) | 7 (7)
access failure (Surgical and medical procedures) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 4 (4)
bowel ischemia (Gastrointestinal disorders) | 3 (3)
thrombosis (Vascular disorders) | 3 (3)
lymphocele (Skin and subcutaneous tissue disorders) | 4 (4)
angina (Cardiac disorders) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm - Placement of TAG Device (N=100)
aortic diameter enlargement (Vascular disorders) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No